CLINICAL TRIAL: NCT04911829
Title: DepressionForefront: Costs, Treatment and Change Process for Dysthymia
Brief Title: Dysthymia: Associated Costs, Treatment and Change Process
Acronym: DFront
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Depression Forefront
Record Dates: First submitted 2017-05-15; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Depression; Cost Benefit Analysis; Psychotherapeutic Processes
Keywords: Dysthymia; Persistent depressive disorder; Chronic depression; Recurrent depression
MeSH Terms: conditions — Depression; Dysthymic Disorder | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inpatient treatment (Active Comparator): High intensity high dosage inpatient short-term psychodynamic psychotherapy
  Interventions: Behavioral: Psychotherapy
- Outpatient treatment (Experimental): Low dosage outpatient short-term psychodynamic psychotherapy
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy

SUMMARY:
The study evaluates cost and effect of inpatient versus outpatient treatment of dysthymia, as well as investigates the processes through which psychotherapy works in treating dysthymia.

DETAILED DESCRIPTION:
Inpatient treatment allows a more intensive treatment and allows the patient to be in a context where it is possible to focus on the processes in therapy with minimal interruption. Outpatient treatment is much less intensive but allows the treatment process to unfold in the context where the patient is experiencing the problems that brought them to therapy. It is not clear which of the contexts will be more effective in alleviating symptoms of dysthymia. Further, as dysthymia is a very costly disease for society it is of interest to know if the two treatments are cost-effective, and which one is the most cost effective.

A great paucity on dysthymia research ha left the psychotherapy field without an understanding of the processes through which dysthymia is changed. This study will investigate the change process through frequent assessments of common factors, psychological processes, symptoms, heart rate variability and cognitive attention bias.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be liberal and similar to clinical practice criteria at the treatment site: Persistent depressive disorder as defined by the diagnostic and statistical manual of mental disorders (DSM5); which includes an International classification of disorders-10 (ICD-10) diagnosis of depression, dysthymia, recurrent depression. unsuccessful previous treatments. living within driving distance from the treatment facilities.

Exclusion Criteria:

* current suicidal risk, current psychosis, marked emotional instability (i.e. issues with impulsivity), strong paranoid traits, current problems related to heavy substance abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive symptoms | At assessment, start (12 weeks after assessment) and end (24 weeks after assessment) of therapy, and at one-year follow up (76 weeks after assessment).
  Beck depression inventory
Change in Depressive symptoms | Once every week for the 12 weeks of active psychotherapy
  Patient health questionnaire
Change in Cost of living with dysthymia | pre therapy, one-year and 10 years
  cost of living with dysthymia, cost-effectiveness of therapy at one-year and at 10 years. Information will be gathered from various registries and combined to a sum of money.

SECONDARY OUTCOMES:
Emotional psychological processes | Once every week for the 12 weeks of active psychotherapy
  weekly measures of central emotional psychological processes (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, lower is better).
cognitive psychological processes | Once every week for the 12 weeks of active psychotherapy
  weekly measures of central cognitive psychological processes (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, lower is better).
metacognitive psychological processes | Once every week for the 12 weeks of active psychotherapy
  weekly measures of central metacognitive psychological processes (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, lower is better).
Common factors-alliance | Once every week for the 12 weeks of active psychotherapy
  weekly measures of central common factors (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, higher is better).
Common factors-expectations | Once every week for the 12 weeks of active psychotherapy
  weekly measures of central common factors (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, higher is better).
Common factors-credibility | Once every week for the 12 weeks of active psychotherapy
  weekly measures of central common factors (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, higher is better).
Common factors-explanation | Once every week for the 12 weeks of active psychotherapy
  weekly measures of central common factors (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, higher is better).
anxiety Symptoms | Once every week for the 12 weeks of active psychotherapy
  weekly measures of Generalized Anxiety Disorders 7-item (GAD7)
resilience | Once every week for the 12 weeks of active psychotherapy
  weekly measures of resilience (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, higher is better).
loneliness | Once every week for the 12 weeks of active psychotherapy
  weekly measures of loneliness (Modum Process Outcome questionnaire, M-poq. Calculated as mean of scores. Range 1-7, higher is better).
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) | Once every week for the 12 weeks of active psychotherapy
  weekly measures of wellbeing. 14 Items scored 1-5 (Total score from 14-70). Higher score is better

CONTACTS AND LOCATIONS:
Overall Officials: Pål Ulvenes, PhD, Principal Investigator — Modum Bad
Locations (1):
- Modum Bad, Vikersund, Buskerud, Norway